CLINICAL TRIAL: NCT00063804
Title: A Phase 1, Dose-Rising Study of AMD11070 in HIV-Seronegative Men to Assess the Safety and Pharmacokinetics After Single or Multiple Doses
Brief Title: Safety of AMD070 When Administered Alone or Boosted With Low-Dose Ritonavir in HIV Uninfected Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5191; 10012 (Registry Identifier: DAIDS ES); ACTG A5191
Record Dates: First submitted 2003-07-07; First posted 2003-07-08 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; CXCR4; AMD11070
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; mavorixafor

ARMS (3):
- 1 (Experimental): escalating single doses of AMD070 ranging from 1/4 to 1 times the maximum tolerated dose (MTD)
  Interventions: Drug: AMD070
- 2 (Experimental): single dose of 200 mg AMD070 after eating a standardized meal
  Interventions: Drug: AMD070
- 3 (Experimental): single dose of 200 mg AMD070 on Days 1, 3, and 17 and single dose of 100 mg ritonavir on Days 3 through 18
  Interventions: Drug: Ritonavir; Drug: AMD070

INTERVENTIONS:
Drug: Ritonavir
  Arms: 3
Drug: AMD070

SUMMARY:
Most currently approved anti-HIV drugs work by stopping the replication of HIV after it has entered cells. AMD070 (also known as AMD11070) is designed to block HIV from entering cells and may be effective in treating patients who have developed resistance to or are unable to take other anti-HIV drugs. This study will evaluate the safety of different doses of AMD070 along with AMD070 boosted with ritonavir (RTV) in HIV uninfected men.

DETAILED DESCRIPTION:
Current therapy for HIV infection primarily uses drugs that inhibit HIV replication via inhibition of viral protease and reverse transcriptase. Many patients either do not tolerate these medications well or develop virologic failure due to incomplete viral suppression and development of antiviral resistance. New drugs target HIV entry into the cell. AMD070 binds to the chemokine receptor CXCR4, inhibiting membrane fusion and viral entry. Animal studies have shown AMD070 to be generally safe and well tolerated. The dose-escalation and drug-drug interaction study will evaluate the safety, tolerability, and pharmacokinetics of single, multiple, and RTV-boosted doses of AMD070 in healthy, HIV uninfected male volunteers.

Participants in this study will be assigned to a single- or multiple-dose AMD070 group (Group 1), a single-dose AMD070 group (Group 2), or an RTV-boosted, multiple-dose AMD070 group (Group 3). Some participants in Group 1 will be given AMD070 once on an empty stomach with no food or drink except for water for 2 hours before and 1 hour after receiving the drug. Up to 4 different doses will be tested in subgroups of Group 1 participants. Some participants in Group 1 will be given AMD070 7 times, 12 hours apart, after eating a standardized breakfast 30 minutes before receiving the drug; 3 different doses will be tested in this group. Participants in Group 2 will be given a single dose of AMD070 after eating a standardized meal. Participants in Group 3 will be given a morning dose of AMD070 on Days 1, 3, and 17 after eating a standardized breakfast 30 minutes before receiving the drug, and a morning and evening dose of RTV on Days 3 through 18. Group 3 participants may also be asked to enroll in an additional study group that will receive a single dose of AMD070 on Days 1 and 3 while fasting.

All participants will be observed as hospital inpatients. Group 1 and 2 participants will stay in the hospital for 24 hours; Group 3 participants will stay in the hospital for 4 days. All participants will have blood and urine collection throughout their hospital stay. Group 3 participants selected to join in the additional study group will have blood and urine samples collected throughout the 5-day study. These participants will be discharged from the hospital on Day 5 and have a follow-up visit around Day 35. All study participants will also undergo an ophthalmologic evaluation and questionnaire sometime after receiving AMD070.

ELIGIBILITY:
Inclusion Criteria for all participants:

* HIV uninfected males in good general health
* Normal electrocardiogram (EKG) and lab values
* Body weight within 33% of ideal weight for height within 28 days of study entry
* Willing to refrain from exercise for 24 hours prior to study entry
* Willing to use acceptable forms of contraception

Inclusion Criteria for Group 3's Additional Study:

* Willing to refrain from consumption of alcohol and grapefruit juice for the duration of the study

Exclusion Criteria for all participants:

* Prescription medications, herbal supplements, or aspirin within 7 days of study entry
* Nonsteroidal anti-inflammatory drugs, over-the-counter medications, and other supplements (including multivitamins) within 1 day of study entry
* Active infection or acute illness within 14 days of study entry
* Drug or alcohol abuse or dependence
* Known sensitivity to AMD070
* History of gastrointestinal bleeding or ulcer
* Any medical or psychological condition that, in the opinion of the investigator, would interfere with study participation

Exclusion Criteria for Group 3:

* Immunizations within 30 days of study entry
* Radiation therapy, cytotoxic chemotherapeutic agents, or immunomodulating agents within 30 days of study entry
* Chronic diarrhea for more than 4 weeks prior to study entry
* Heart conduction abnormalities, heart arrhythmias, cardiomyopathy, any repolarization delay, or other risk factors for heart failure and hypokalemia

Exclusion Criteria for Group 3's Additional Study:

* Grade 3 or 4 adverse event while participating in Group 3
* Consumption of alcohol within 48 hours of study entry

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
AMD070 pharmacokinetic (PK) parameters under three conditions, and the within-volunteer differences between them
Steady-state RTV PK parameters
Grade 3 and 4 adverse effects, as defined by the protocol

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hendrix, MD, Study Chair — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] De Clercq E. HIV-chemotherapy and -prophylaxis: new drugs, leads and approaches. Int J Biochem Cell Biol. 2004 Sep;36(9):1800-22. doi: 10.1016/j.biocel.2004.02.015. PMID 15183346
- [Background] Marks K, Gulick RM. New antiretroviral agents for the treatment of HIV infection. Curr HIV/AIDS Rep. 2004 Jun;1(2):82-8. doi: 10.1007/s11904-004-0012-0. PMID 16091227
- [Background] Princen K, Schols D. HIV chemokine receptor inhibitors as novel anti-HIV drugs. Cytokine Growth Factor Rev. 2005 Dec;16(6):659-77. doi: 10.1016/j.cytogfr.2005.05.009. Epub 2005 Jul 6. PMID 16005254
- [Background] Schols D. HIV co-receptors as targets for antiviral therapy. Curr Top Med Chem. 2004;4(9):883-93. doi: 10.2174/1568026043388501. PMID 15134547
- [Result] Stone ND, Dunaway SB, Flexner C, Tierney C, Calandra GB, Becker S, Cao YJ, Wiggins IP, Conley J, MacFarland RT, Park JG, Lalama C, Snyder S, Kallungal B, Klingman KL, Hendrix CW. Multiple-dose escalation study of the safety, pharmacokinetics, and biologic activity of oral AMD070, a selective CXCR4 receptor inhibitor, in human subjects. Antimicrob Agents Chemother. 2007 Jul;51(7):2351-8. doi: 10.1128/AAC.00013-07. Epub 2007 Apr 23. PMID 17452489
- [Result] Cao YJ, Flexner CW, Dunaway S, Park JG, Klingman K, Wiggins I, Conley J, Radebaugh C, Kashuba AD, MacFarland R, Becker S, Hendrix CW. Effect of low-dose ritonavir on the pharmacokinetics of the CXCR4 antagonist AMD070 in healthy volunteers. Antimicrob Agents Chemother. 2008 May;52(5):1630-4. doi: 10.1128/AAC.01460-07. Epub 2008 Feb 19. PMID 18285477